CLINICAL TRIAL: NCT05768763
Title: SEARCH Multisectoral Strategy to Address Persistent Drivers of the HIV Epidemic in East Africa Phase B
Brief Title: SEARCH SAPPHIRE Phase B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Infectious Diseases Research Collaboration, Uganda (Other); Makerere University (Other); Kenya Medical Research Institute (Other); University of California, Berkeley (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institute of Mental Health (NIMH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SEARCH SAPPHIRE Phase B; U01AI150510 (NIH)
Record Dates: First submitted 2023-03-03; First posted 2023-03-14 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: HIV
Keywords: PrEP; HIV Treatment; HIV Prevention; Community Health; Youth and Adolescents; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: In the "evaluation" Phase B, the SEARCH SAPPHIRE study will evaluate the effects of Dynamic Prevention and Dynamic Treatment intervention packages based on data from Phase A (NCT04810650) and new advances from outside the study delivered in a precision community health model, on HIV incidence and other health outcomes, in a pair-matched community randomized design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precision Community Health (Experimental): The Phase B precision community health intervention will consist of a three part intervention: 1) Community-enhanced reach activities 2) Person-centered care delivery; and, 3) Data system enhancement to improve reach and person-centered delivery
  Interventions: Behavioral: Community-enhanced reach activities; Behavioral: Person-centered care delivery; Other: Data system enhancement to improve reach and person-centered delivery
- Control (Active Comparator): Standard of Care
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Community-enhanced reach activities — We will conduct a series of community engagement activities designed to reach persons at risk for HIV, undiagnosed with HIV or diagnosed, or hypertension, and fallen out of care, working closely with community health workers, integrated in the community health system.
  Arms: Precision Community Health
Behavioral: Person-centered care delivery — Structured approach to provide patient-centered biomedical options for HIV prevention (dynamic choice prevention). Tailored services for HIV treatment support using structured life stage evaluation and assessment plan (LEAP) for youth, pregnant women, and persons with or at risk of HIV viral non-suppression, that includes counselling for heavy alcohol users. Structured approach to offer telehealth for severe hypertension follow up.
  Arms: Precision Community Health
Other: Data system enhancement to improve reach and person-centered delivery — Both community-enhanced reach and person-centered delivery will be strengthened through a customized in-country Ministry of Health-compatible community health worker smartphone app and two-way data system linking community health workers and clinical records.
  Arms: Precision Community Health
Behavioral: Standard of Care — Standard of Care in Uganda and Kenya
  Arms: Control

SUMMARY:
This study will evaluate the effects of optimized dynamic prevention and treatment packages delivered in a precision community health model on HIV incidence, as well as other health outcomes, in a community randomized trial design.

DETAILED DESCRIPTION:
In the "evaluation" Phase B, the SEARCH SAPPHIRE study will evaluate the effects of Dynamic Prevention and Dynamic Treatment intervention packages based on data from Phase A (NCT04810650) and new advances from outside the study delivered in a precision community health model, on HIV incidence and other health outcomes, in a pair-matched community randomized design.

The Phase B precision community health intervention will consist of a three part intervention: 1) Community-enhanced reach activities 2) Person-centered care delivery; and, 3) Data-enhancement to improve precision of interventions.

The study hypothesis for the Phase B population level study is: A Precision Community Health Model leveraging existing facility-based outreach and community health workers, enabled by dynamic choice prevention/treatment multi-disease approaches and interactive data systems -will reduce HIV infections, deaths and improve health.

Structured stakeholder consultations are formally incorporated in the study design and leverage regular and ongoing collaborations the study team has with the HIV, non-communicable disease and general health leads in Kenya and Uganda Ministries of Health and PEPFAR implementing partners at the national and the regional level.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 15 years
2. Living in SEARCH study communities
3. Provided informed consent

Exclusion Criteria:

1. <15 years of age
2. Living outside SEARCH study communities
3. Unable to provide consent or parental co-consent as per country guidelines

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80000 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
HIV incidence | 24 months
  HIV incidence per 100 person-year

SECONDARY OUTCOMES:
Population-Level Viremia | 24 months
  Proportion of adults with plasma RNA levels > 1000 c/mL
Prevention Coverage | assessed between 18-24 month follow up
  Proportion of HIV-negative follow-up months during which PrEP/PEP was used
Population Level Viral Suppression among PWH | assessed between 18-24 month follow up
  Proportion of HIV+ adults with plasma RNA level <400 cps/mL
Mortality risk | assessed between 18-24 month follow up
  Mortality risk of all community members aged ≥ 15 years at baseline
Hypertension Control | assessed between 18-24 month follow up
  HTN control (BP <140/90 mmHG) of community members aged ≥ 40 years with blood pressure >160/100 mmHG
Severe Hypertension | assessed between 18-24 month follow up
  Severe HTN (BP >160/100 mmHG)
Persons presenting with late HIV disease | assessed between 18-24 month follow up
  Proportion of PWH adults with CD4 T-cell count < 200
Late Pediatric HIV Diagnosis | assessed between 18-24 month follow up
  Proportion of children of HIV+/unknown status mothers diagnosed with HIV
Heavy Alcohol Use | assessed between 18-24 month follow up
  AUDIT-C score ≥3 for women, ≥4 for men
HPV Immunization Coverage | assessed between 18-24 month follow up
  Proportion of adolescent girls who have received ≥1 HPV vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Diane Havlir, MD, Principal Investigator — University of California, San Francisco; Moses Kamya, MBChB, PhD, Principal Investigator — Makerere University; Infectious Diseases Research Collaboration; Maya Petersen, PhD, Principal Investigator — University of California, Berkeley
Locations (2):
- SEARCH Office / GPRT, Kisumu, Kenya
- Infectious Diseases Research Collaboration, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No